CLINICAL TRIAL: NCT06042725
Title: Phase I Clinical Trial of Bcl2 Inhibitor Venetoclax in Combination With Lenalidomide and Dexamethasone (Ven-Rd), Daratumumab and Dexamethasone (Ven-Dd), or Daratumumab-Lenalidomide-Dexamethasone (Ven-DRd) in t(11;14) Multiple Myeloma
Brief Title: MC210808 Venetoclax in Combination With Lenalidomide and Dexamethasone (Ven-Rd), Daratumumab and Dexamethasone (Ven-Dd), or Daratumumab-Lenalidomide-Dexamethasone (Ven-DRd) for the Treatment of Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC210808; NCI-2023-06776 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC210808 (Other: Mayo Clinic in Rochester); 22-009930 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-09-12; First posted 2023-09-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Biopsy; X-Rays; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; Magnetic Resonance Spectroscopy; venetoclax; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Ven-Dd) (Experimental): Patients receive venetoclax PO QD on days 1-28 of each cycle, daratumumab SC on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7+, and dexamethasone PO on days 1, 8, 15, 22 of cycles 1-12. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo chest x-ray and optional collection of blood samples during screening. In addition, patients undergo x-rays, WBLDCT, PET/CT or MRI scans during screening and on study, and bone marrow aspiration and biopsy during screening, and during follow-up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Chest Radiography; Procedure: Computed Tomography; Biological: Daratumumab; Drug: Dexamethasone; Procedure: Low Dose Computed Tomography of the Whole Body; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Venetoclax; Procedure: X-Ray Imaging; Other: Questionnaire Administration
- Arm B (Ven-Rd) (Experimental): Patients receive venetoclax PO QD on days 1-28 of each cycle, lenalidomide PO QD on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, 22 of cycles 1-12. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo chest x-ray and optional collection of blood samples during screening. In addition, patients undergo x-rays, WBLDCT, PET/CT or MRI scans during screening and on study, and bone marrow aspiration and biopsy during screening, and during follow-up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Chest Radiography; Procedure: Computed Tomography; Drug: Dexamethasone; Drug: Lenalidomide; Procedure: Low Dose Computed Tomography of the Whole Body; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Venetoclax; Procedure: X-Ray Imaging; Other: Questionnaire Administration
- Arm C (Ven-DRd) (Experimental): Patients receive venetoclax PO QD on days 1-28 of each cycle, daratumumab SC on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7+, lenalidomide PO QD on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of cycles 1-12. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo chest x-ray and optional collection of blood samples during screening. In addition, patients undergo x-rays, WBLDCT, PET/CT or MRI scans during screening and on study, and bone marrow aspiration and biopsy during screening, on study, and during follow-up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Chest Radiography; Procedure: Computed Tomography; Biological: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Procedure: Low Dose Computed Tomography of the Whole Body; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Venetoclax; Procedure: X-Ray Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo optional collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Daratumumab — Given SC
  Other Names: 945721-28-8; Daratumumab Biosimilar HLX15; Daratumumab-fihj; Darzalex; HLX15; HuMax-CD38; JNJ-54767414
  Arms: Arm A (Ven-Dd); Arm C (Ven-DRd)
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm B (Ven-Rd); Arm C (Ven-DRd)
Procedure: Low Dose Computed Tomography of the Whole Body — Undergo WBLDCT
  Other Names: Low-dose Whole-body CT; Whole Body Low Dose Computed Tomography; Whole Body Low Dose CT; Whole-body Low-dose CT
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Procedure: X-Ray Imaging — Undergo x-rays
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of venetoclax in combination with lenalidomide and dexamethasone, daratumumab and dexamethasone, or daratumumab, lenalidomide, and dexamethasone in treating patients with multiple myeloma. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Lenalidomide is a drug that is similar to thalidomide, and is used to treat multiple myeloma and certain types of anemia. Lenalidomide belongs to the family of drugs called angiogenesis inhibitors. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Daratumumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD38, which is found on some types of immune cells and cancer cells, including myeloma cells. Daratumumab may block CD38 and help the immune system kill cancer cells. Adding venetoclax to the other drug combinations may allow control of the cancer than is possible with the current treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the recommended phase II dose (RP2D) of venetoclax that can be combined with standard dose daratumumab and dexamethasone (Dd) (Arm A), lenalidomide and dexamethasone (Rd) (Arm B) or daratumumab, lenalidomide and dexamethasone (DRd) (Arm C) in patients with t(11;14) multiple myeloma (MM).

SECONDARY OBJECTIVES:

I. To assess frequency and severity of treatment-emergent adverse events (TEAEs) graded per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

II. To assess best response while on treatment per International Myeloma Working Group (IMWG) criteria.

EXPLORATORY OBJECTIVE:

I. To examine the effect of treatment on patient reported toxicity and quality of life using validated tools.

OUTLINE: This is a dose-escalation study of venetoclax. Patients with relapsed MM (Group 1) are assigned to Arm B or C. Patients with newly diagnosed MM (Group 2) are assigned to Arm A, B, or C.

ARM A: Patients receive venetoclax orally (PO) once daily (QD) on days 1-28 of each cycle, daratumumab subcutaneously (SC) on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7+, and dexamethasone PO on days 1, 8, 15, 22 of cycles 1-12. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo chest x-ray and optional collection of blood samples during screening. In addition, patients undergo x-rays, whole-body low-dose computed tomography (WBLDCT), positron emission tomography (PET)/computed tomography (CT) or magnetic resonance imaging (MRI) scans during screening and on study, and bone marrow aspiration and biopsy during screening, and during follow-up

ARM B: Patients receive venetoclax PO QD on days 1-28 of each cycle, lenalidomide PO QD on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, 22 of cycles 1-12. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo chest x-ray and optional collection of blood samples during screening. In addition, patients undergo x-rays, WBLDCT, PET/CT or MRI scans during screening and on study, and bone marrow aspiration and biopsy during screening, and during follow-up.

ARM C: Patients receive venetoclax PO QD on days 1-28 of each cycle, daratumumab SC on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7+, lenalidomide PO QD on days 1-21 of each cycle, and dexamethasone PO on days 1, 8, 15, and 22 of cycles 1-12. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo chest x-ray and optional collection of blood samples during screening. In addition, patients undergo x-rays, WBLDCT, PET/CT or MRI scans during screening and on study, and bone marrow aspiration and biopsy during screening, on study, and during follow-up.

After completion of study treatment, patients are followed up at 30 days and then every 3 or 6 months for a total of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Diagnosis of active MM with bone marrow plasma cell fluorescence in situ hybridization (FISH) test run under an Investigational Device Exemption (IDE) demonstrating of t(11;14), either from time of diagnosis or confirmed with IDE at Mayo Clinic after time of diagnosis, during screening period for study. Note: Samples tested beyond 72 hours from the collection will not be considered adequate for trial enrollment
* PRE-REGISTRATION: Group 1 - At least one prior line of therapy which did not include venetoclax
* PRE-REGISTRATION: Group 2 - No more than 1 cycle of any commonly used myeloma regimen for treatment of newly diagnosed MM
* PRE-REGISTRATION: Patient is not being considered for stem cell transplant (group 2, newly diagnosed only)
* REGISTRATION: Age ≥ 18 years
* REGISTRATION: Calculated creatinine clearance (using Cockcroft-Gault equation) ≥ 30 mL/min (obtained ≤ 14 days prior to registration)
* REGISTRATION: Absolute neutrophil count (ANC) ≥ 1000/uL (without growth factor support) (obtained ≤ 14 days prior to registration)
* REGISTRATION: Un-transfused Platelet count ≥ 75000/uL (≥ 50,000/uL if marrow plasma cells [PC]% > 50%) (obtained ≤ 14 days prior to registration)
* REGISTRATION: Hemoglobin ≥ 8.0 g/dL (transfusion permitted) (obtained ≤ 14 days prior to registration)
* REGISTRATION: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (known Gilbert's syndrome are allowed provided bilirubin ≤ 2.5 mg/dL) (obtained ≤ 14 days prior to registration)
* REGISTRATION: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (obtained ≤ 14 days prior to registration)
* REGISTRATION: Alkaline phosphatase ≤ 750 U/L (obtained ≤ 14 days prior to registration)
* REGISTRATION: Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein ≥ 1.0 g/dL
  * ≥ 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* REGISTRATION: Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* REGISTRATION: Provide written informed consent
* REGISTRATION: Ability to complete questionnaire(s) by themselves or with assistance
* REGISTRATION: Negative serum pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only
* REGISTRATION: Willing to follow strict birth control measures as suggested by the study
* REGISTRATION: Female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP) OR
  * Due to lenalidomide being a thalidomide analogue with risk for embryo-fetal toxicity and prescribed under a pregnancy prevention/controlled distribution program, WOCBP participants will be eligible if they commit to either:

    * Abstain continuously from heterosexual sexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
    * To use birth control as follows:

      * Two methods of reliable birth control (one method that is highly effective and one additional effective (barrier) method), beginning 4 weeks prior to initiating treatment with lenalidomide, during therapy, during dose interruptions and continuing for 4 weeks following discontinuation of lenalidomide treatment
* REGISTRATION: Male participants are eligible to participate if they agree to the following from the time of first dose of study treatment until 28-days after the last dose of lenalidomide, to allow for clearance of any altered sperm:

  * Refrain from donating sperm PLUS either:

    * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
    * Must agree to use contraception/barrier as detailed below:

      * Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of < 1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females)
* REGISTRATION: Life expectancy ≥ 12 weeks
* REGISTRATION: Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* REGISTRATION: Willing to provide research bone marrow aspirate specimen
* REGISTRATION: Willing to follow the requirements of the Revlimid (Registered Trademark) Risk Evaluation and Mitigation Strategy (REMS) program. Note: Exception for Group 2 patients enrolled on Arm A

Exclusion Criteria:

* PRE-REGISTRATION: History of any active malignancy within the past 2 years prior to screening, with the exception of:

  * Adequately treated carcinoma in situ of the uterine cervix
  * Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin
  * Asymptomatic prostate cancer with no requirement for therapy
  * Previous malignancy surgically resected (or treated with other modalities) with curative intent
* REGISTRATION: Other concurrent chemotherapy or any ancillary therapy considered investigational

  * Note: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* REGISTRATION: Major surgery ≤ 14 days prior to study registration
* REGISTRATION: History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* REGISTRATION: Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* REGISTRATION: Administration of strong/moderate CYP3A inhibitors or inducers ≤ 28 days prior to registration
* REGISTRATION: Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* REGISTRATION: Participation in other clinical trials, including those with other investigational agents not included in this trial, ≤ 30 days prior to registration
* REGISTRATION: Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of venetoclax including difficulty swallowing REGISTRATION: Heart failure > New York Heart Association (NYHA) class II
* REGISTRATION: Presence of positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment

  * Note: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative hepatitis C RNA test is obtained
  * Note: Hepatitis RNA testing is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 28 Days (1 treatment cycle); Up to 3 years
  Dose-limiting toxicities (DLT) are defined according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events | Up to 30 days after completion of study treatment
  The number and severity of all adverse events (overall and by dose- level) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion. This will provide an indication of the level of tolerance for this treatment combination in this patient group.
Best response while on treatment | Up to 3 years
  The overall response rate and ≥ very good partial response (VGPR) rate will be estimated by the number of patients with each response category (e.g., stringent complete response, complete response, VGPR, partial response, etc) divided by the total number of evaluable patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials